CLINICAL TRIAL: NCT05106504
Title: Effect of Medical Cannabis for Non-motor Symptoms of Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Saar Anis, Principal investigator. Senior Neurologist, Movement Disorders Institute, Sheba Medical Center, Sheba Medical Center
Other Study IDs: Sheba-20-7553-SA-CTL
Record Dates: First submitted 2021-10-16; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Bladder, Overactive; Parkinson Disease
Keywords: non-motor symptoms; Parkinson's disease; Bladder overactivity; Medical cannabis; Cannabidiol; delta-9-tetrahydrocannabinol; pain
MeSH Terms: conditions — Urinary Bladder, Overactive; Parkinson Disease; Pain | interventions — Medical Marijuana

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's disease patients: Parkinson's disease patients receiving medical cannabis for pain related to the disease
  Interventions: Drug: Medical Cannabis

INTERVENTIONS:
Drug: Medical Cannabis — Patients will be assessed before and after use of Medical cannabis via inhaled dried buds or sublingual oil extract

SUMMARY:
Medical cannabis (MC) is a standard treatment in Israel to Parkinson's disease (PD) patients suffering from pain. Nevertheless, it is not known about MC effectiveness for other non-motor symptoms of the disease. Our aim is to prospectively observe patients with PD before and after initiation of MC, for non-motor symptoms effect. In specific, relying of data from multiple sclerosis patients and basic science showing cannabinoid receptor 1 (CB1) is abundantly expressed in the sub epithelial layer of the bladder, we will explore the impact of MC on bladder function and urinary symptoms.

DETAILED DESCRIPTION:
This is a prospective, open-label, observational study. Patients with Parkinson's disease (PD) receiving licensure from Israeli Ministry of Health (MOH) for using medical cannabis (MC) for PD related symptoms and pain, being followed up in the Movement Disorders Institute (MDI) at SHEBA Medical Center (SMC) will be eligible to participate. Assessment regarding patient demographic, disease characteristics (Hoehn and Yahr, disease duration, disease first symptom etc.) will be collected at baseline along with designated questionnaires to evaluate the non-motor symptoms (NMSS, PDSS, Kings PD pain scale, PDQ8) and urinary function (Bladder over activity, International prostate symptom score (IPSS) and nocturia questionnaires). after MC initiation, patients will be observed and evaluated for the impact of MC 4-8 weeks following treatment initiation. Also, for each patient, MC being used will be analyzed in order to expose relationship between phyto-cannabinoid content and efficacy or side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease according to UK Parkinson's disease society barin bank clinical diagnostic criteria
* Holds a validated Medical cannabis license, from Israeli Ministry of health
* Able to sign informed consent
* Age 18-80

Exclusion Criteria:

* Use of Medical cannabis in the previous 30 days prior to study recruitment visit
* Concomitent severe co-morbidities able to influence outcomes such as spinal injury, cancer, dementia.
* Cannot sign informed consent

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Current study population include PD patients, males and females, aged 18-80, with a license to use Medical cannabis for PD related symptoms, newly issued or, with no recent use.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change in Non-motor symptoms scale (NMSS) | before and 4-8 weeks after treatment initiation
  NMSS will be assessed before and after medical cannabis use, range 0-360, higher scores mean a worse outcome
Change in Bladder over activity symptoms | before and 4-8 weeks after treatment initiation
  Overactive Bladder Symptom Score (OABSS) questionnaires will be assessed before and after medical cannabis use, range 0-15, higher scores mean a worse outcome

SECONDARY OUTCOMES:
Change in sleep quality | before and 4-8 weeks after treatment initiation
  PDSS questionnaire will be employed before and after MC use, range 0-28, higher scores mean a worse outcome
Change in subjective Pain | before and 4-8 weeks after treatment initiation
  Kings PD pain scale will be employed before and after MC use, range 0-168 , higher scores mean a worse outcome
Change in Quality of life | before and 4-8 weeks after treatment initiation
  PDQ8 questionnaire will be employed before and after MC use, range 0-32 , higher scores mean a worse outcome
Cannabis strand analysis | 4-8 weeks following treatment initiation
  Cannabinoid content within products being used by our patient will be analyzed. Correlation between efficacy and side effect profile to MC cannabinoid content will be employed
Change in International prostate symptom score (IPSS) | before and 4-8 weeks after treatment initiation
  IPSS will be assessed before and after medical cannabis use, range 0-35, higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Saar Anis, MD, Principal Investigator — Sheba Medical Center, Ramat-Gan, Israel
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No